CLINICAL TRIAL: NCT04061148
Title: Clinical Testing of Near Infrared Spectroscopy (NIRS) for Quantitative Assessment of Depression
Brief Title: Near Infrared Spectroscopy (NIRS) for Assessment of Depression
Acronym: NIRSIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: OBELAB, Inc. (Industry); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-22188
Record Dates: First submitted 2019-02-20; First posted 2019-08-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
Keywords: Near Infrared Spectroscopy; Depression; NIRS; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Repeated NIRS measure comparison of patients being treated for Major Depressive Disorder with control, non-depressed subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Non-Depressed Controls (Other): Volunteers who have screened by a clinical psychiatrist, to exclude depression and other major psychiatric and neurocognitive disorders.
  They will undergo NIRSIT testing to measure frontal blood oxygenation up to 3 times, with an interval of 3 weeks between each measurement.
  Interventions: Device: NIRSIT
- Depressed Patients (Active Comparator): Patients diagnosed with Major Depressive Disorder by a clinical psychiatrist. They will undergo NIRSIT testing to measure frontal blood oxygenation up to 5 times, with an interval of 3 weeks between each measurement, over the course of their clinical therapy for Major Depressive Disorder.
  Interventions: Device: NIRSIT

INTERVENTIONS:
Device: NIRSIT — NIRSIT is a device that utilizes Near Infrared Spectroscopy to provide a non-invasive measurement of frontal lobe blood oxygenation over time.

SUMMARY:
Develop a NIRSIT testing protocol that can be administered in the diagnostic setting and reliably distinguishes the symptoms and severity of depression, with the help of repeated measure (up to five visits per subject) comparison of patients being treated for Major Depressive Disorder with control, non-depressed subjects.

DETAILED DESCRIPTION:
Background & Significance:

The history of utilizing the near infrared (NIR) spectrum (650-1000nm) in cognitive studies is chronicled in a recent review. Taking advantage of the facts that human tissue is relatively transparent to NIR and hemoglobin absorbs those wavelengths of light, in 1977, Jobsis developed a non-invasive device able to detect oxygenation changes in the brain. He later used this technique to study cerebral oxygenation in new born infants. The first publications describing NIRS results began to appear in the early 1990s, and in 2000, the first commercially available device was marketed. In 2009, Hitachi released the first battery operated wireless/ wearable device. In the 3 years preceding this 2012 review, ~400 articles utilizing this technology have been published in the fields of neurology (Alzheimer's disease, dementia, depression, epilepsy, Parkinson's, rehabilitation, stroke), psychiatry (anxiety, substance abuse, schizophrenia), education (attention, comprehension, reasoning) and basic research (pain, sleep).

Device:

Near Infrared Spectroscopy (NIRS) provides a non-invasive measurement of frontal lobe blood flow and saturation over time. The NIRSIT device has ninety-six (96) two color infrared lasers and paired photodiodes which record oxygen saturation to a depth of 2 cm from the frontal cortex of humans. NIRSIT provides a measurement of blood saturation from over 200 prefrontal regions providing high spatial resolution at a scan rate of 32 Hz providing high temporal resolution. NIRSIT can provide real-time cognitive studies which can discriminate cognitive workload, concentration, and emotional stress and anxiety. NIRS provides 200 measurements of oxy, deoxy, total hemoglobin, and heart rate 32 times per second.

Non-Significant Risk Justification:

No clinical decisions will be made based on the data acquired for this study. The NIRSIT data is collected solely for the study. The NIRSIT data will not be used for any clinical decision making and therefore the study qualifies for NSR.

NIRS has been studied in Japan since 20001. The OBE Lab NIRSIT device has more sensors than the Hitachi ETG-4000, which has US 510K clearance (K042501) since Oct 12 2004 with an intended use of the measurement of relative levels of cerebral deoxyhemoglobin and oxyhemoglobin, but has a similar safety profile. The OBE Lab NIRSIT device has a higher sensor count (96), higher number of assessed voxels (200), higher temporal resolution (30 Hz), but similar safety profile to the Hitachi ETG-4000. The Hitachi ETG-4000 would be the predicate device for FDA 510K clearance.

Methods:

On the day of NIRSIT testing, depressive symptoms of subjects will be measured using the Hamilton B Depression Rating Scale (HDRS), the Beck Depression Index (BDI) and Patient Health Questionnaire-9 (PHQ-9), and a cognitive assessment (Mini International Neuropsychiatric interview) will be administered prior to NIRSIT testing. We will take front and side photos of subjects to document how the device was placed.

The cognitive tasks will include cartoon humor reaction test, where subjects will be shown a series of humorous cartoons and verbal fluency task, where they will be asked to say words that begin with certain letters. We will make an audio recording of the words they say, to validate the number of correct words.

Testing sessions will be repeated up to five times depending on the amount of variability when compared to previous sessions with that subject.

Controls will be selected to reflect the age distribution of patients treated at our institution for MDD in the past two years.

Psychiatry collaborators will be informed of survey response that indicates possible suicide ideation.

Sample Size: Control Group - 30 volunteers Control subjects will be SFVAMC patients, staff or general public who self-indicate that they are not depressed.

Patient Group - 60 patients with Major Depressive Disorder MDD patient group will also include those whose initial depressive symptoms were sufficiently severe such that they and their treating physician have decided that they may benefit from treatments such as electroconvulsive therapy (ECT) or ketamine infusion.

Recruitment: For the healthy controls, a flyer describing the study will be posted outside the Anesthesia Business Office, at the San Francisco VA Medical Center. One of the study clinical attendings will administer the MINI (Mini International Neuropsychiatric Interview) test to ensure that the controls do not have any conditions that would exclude them from participating in the study.

Patients will be identified and approached by study Psychiatrists and asked if they would like to participate in the study. They will be given a flyer that explains the study, to improve the consent process. After patients have been screened and have signed the informed consent form to participate in the study, they will be enrolled in the study. One of the study psychiatrists will administer the MINI (Mini International Neuropsychiatric Interview) test to ensure that the patients do not have any conditions that would exclude them from participating in the study.

Informed consent will be obtained by the attending psychiatrist, the principal or coinvestigator

Statistical Methods: Collaborators and colleagues will evaluate the tasks that are available in the NIRSIT software and select which produce the highest readouts and evaluate which channels detect changes prior to enrolling any subjects.

Principal component analysis will be used to determine which channels to focus examination. Previous examinations focused on the bilateral frontopolar area (Broadmann areas [BA] 9 and 46), ventro-lateral (BA 44, 45, 47) and fronto-polar (BA 10)5,10,11.

Rhythmic signals that indicate noise artifacts and body movement artifacts will be removed.

Mean changes in blood flow will be calculated using linear fit between the final 10 s of the pre-task period and the final 5 s of the post-task period.

Test-retest intra-class correlation will be performed at the single-subject level to evaluate the reproducibility of results and indicate whether further testing is indicated for controls and MDD patients during their treatment course.

ANOVA and the F statistic will be used to compare the degree of changes across groups.

Ex-Gaussian modeling will be used to compare response times and misses across severity of depression.

Results will be adjusted for differences in age, the presence of post-traumatic stress disorder (PTSD), substance abuse (drugs or alcohol), suicide history, anxiety, comorbidities including heart, liver or kidney disease, diabetes, cancer and medications including anti-psychotics, antidepressants, anti-anxiety and pain medications.

Risks:

* Loss of privacy. All clinical studies have some risk for loss of privacy. Medical and psychiatric records are reviewed by study staff and recorded for research purposes. All records will be stored as encrypted files or in locked storage to reduce risks.
* NIRSIT device uses infrared light. The FDA has concluded that the light emitted by the device is harmless and poses non-significant risk.

Minimizing Risk:

1. All study records are stored in locked file cabinets in locked offices. The risk of loss of study related materials is small.
2. NIRSIT and depression inventory testing will be done in a manner that is sensitive to patient needs and minimizes possible embarrassment.
3. Patients will be screened for suicidality at each screening visit. Patients who indicate on the BDI or PHQ-9 survey they have thoughts that they would be better off dead or hurting themselves will be brought to the attention of the treating physician. The treating physician will be filling in the HAM-D and will therefore, be investigating suicidal intention as part of standard of care, using a progress note to indicate any further action needed.

Benefits:

NIRSIT and depression inventory testing pose no more than minimal risk to subjects. This study may show that the device and testing protocol are able to improve the sensitivity and specificity of depression diagnostics and thereby make possible more specific treatments and therapy improve the care of future patients with depression.

Qualifications of Investigators:

Dr. Arthur Wallace, M.D., Ph.D. has done medical research since 1978 including large animal, human clinical trials, and human physiological measurement. He has a Ph.D. in biomedical engineering and completed a medical internship, anesthesia residency, and a fellowship in cardiac anesthesiology. He has been a faculty member of anesthesiology at UCSF since 1992 during this time he has been the PI on several clinical trials in high risk patients including the Afterload, Warm Cardioplegia, Atenolol, Clonidine, EDRF Intraop, L-ARG, AVD Study, PCRRT, and Aneurysm Trials. Dr. Wallace has worked with impedance devices since 1991 and has been the chief scientific adviser on the ECOM projects since their inception in 1996, as well as member of VA IACUC. He has been responsible for the tube design, algorithm development, electronic design, in-vivo experiments, as well as the animal and human trials.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who sign informed consent.
* Controls: Volunteers over 18 years of age who are not depressed.
* Patients over 18 years of age with a diagnosis of Major Depressive Disorder, receiving clinical therapy at SFVAMC.

Exclusion Criteria:

* Subjects who cannot sign informed consent.
* Exclusion criteria for control subjects: 1.Depression 2.Anxiety, psychotic, substance abuse, mood and personality disorders 3.Major neurocognitive disorders such as Alzheimer's disease and other dementias 4.Neurologic disorders with anatomic lesions including traumatic brain injury, stroke, tumor and arteriovenous malformation
* Exclusion criteria for depressed patients: 1.Psychotic disorders like schizophrenia 2.Major neurocognitive disorders such as Alzheimer's disease and other dementias 3.Neurologic disorders with anatomic lesions including traumatic brain injury, stroke, tumor and arteriovenous malformation 4.Not receiving clinical therapy for depression at SFVAMC'

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Frontal Oxyhemoglobin concentration before initiation of treatment for MDD | Each measurement is over 10 to 15 mins long, taken during the performance of VFT and CHR, on the day of initiation of treatment for MDD, but before the treatment is given.
  Change in Oxyhemoglobin concentration in frontal blood from the baseline during the performance of Verbal Fluency Task (VFT) and Cartoon humor reaction task (CHR) by the subject.
Change in Frontal Oxyhemoglobin concentration 3 weeks after initiation of treatment for MDD | Each measurement is over 10 to 15 mins long, taken during the performance of VFT and CHR, 3 weeks after initiation of treatment for MDD.
  Change in Oxyhemoglobin concentration in frontal blood from the baseline during the performance of Verbal Fluency Task (VFT) and Cartoon humor reaction task (CHR) by the subject.
Change in Frontal Oxyhemoglobin concentration 6 weeks after initiation of treatment for MDD | Each measurement is over 10 to 15 mins long, taken during the performance of VFT and CHR, 6 weeks after initiation of treatment for MDD.
  Change in Oxyhemoglobin concentration in frontal blood from the baseline during the performance of Verbal Fluency Task (VFT) and Cartoon humor reaction task (CHR) by the subject.
Change in Frontal Deoxyhemoglobin concentration before initiation of treatment for MDD | Each measurement is over 10 to 15 mins long, taken during the performance of VFT and CHR, on the day of initiation of treatment for MDD, but before the treatment is given.
  Change in Deoxyhemoglobin concentration in frontal blood from the baseline during the performance of Verbal Fluency Task and Cartoon humor reaction task by the subject.
Change in Frontal Deoxyhemoglobin concentration 3 weeks after initiation of treatment for MDD | Each measurement is over 10 to 15 mins long, taken during the performance of VFT and CHR, 3 weeks after initiation of treatment for MDD.
  Change in Deoxyhemoglobin concentration in frontal blood from the baseline during the performance of Verbal Fluency Task and Cartoon humor reaction task by the subject.
Change in Frontal Deoxyhemoglobin concentration 6 weeks after initiation of treatment for MDD | Each measurement is over 10 to 15 mins long, taken during the performance of VFT and CHR, 6 weeks after initiation of treatment for MDD.
  Change in Deoxyhemoglobin concentration in frontal blood from the baseline during the performance of Verbal Fluency Task and Cartoon humor reaction task by the subject.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) Score | HAM-D is administered before each of the three NIRS measurement sessions; on the day of initiation of treatment for MDD, but before the treatment is given; 3 weeks after initiation of treatment and 6 weeks after the initiation of treatment.
  Changes in HAM-D Scores before, during and after treatment of MDD. The score range is 0-50, with 50 indicating most severe depression.
Beck's Depression Inventory - II (BDI-II) Scores | BDI-II is administered before each of the three NIRS measurement sessions; on the day of initiation of treatment for MDD, but before the treatment is given; 3 weeks after initiation of treatment and 6 weeks after the initiation of treatment.
  Changes in BDI-II Scores before, during and after treatment of MDD. The score range is 0-63, with 63 indicating most severe depression.
Patient Health Questionnaire-9 (PHQ-9) Scores | PHQ-9 is administered before each of the three NIRS measurement sessions; on the day of initiation of treatment for MDD, but before the treatment is given; 3 weeks after initiation of treatment and 6 weeks after the initiation of treatment.
  Changes in PHQ-9 Scores before, during and after treatment of MDD. The score range is 0-27, with 27 indicating most severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Wallace, MD, PhD, Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT04061148/Prot_001.pdf